CLINICAL TRIAL: NCT01719445
Title: Remote Food Photography for the Real-time Measurement of Children's Food Intake
Brief Title: The Food Phone Project
Acronym: FPP
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 10040; R01DK089051 (NIH)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Comparison of Energy Intake Methods
Keywords: Energy Intake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine collection as part DLW procedure.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- RFPM/Paper and Pen Method

SUMMARY:
The Primary Aim of the project is to modify the RFPM for adolescents and to address the concerns identified by the reviewers of the first grant application. We will then test the RFPM's validity (accuracy) compared to the validity of pen-and-paper food records.

DETAILED DESCRIPTION:
The Primary Aim of the project is to modify the RFPM for adolescents and to address the concerns identified by the reviewers of the first grant application. We will then test the RFPM's validity (accuracy) compared to the validity of pen-and-paper food records. Our experience and the literature indicate that the RFPM is acceptable and feasible in school settings. Following modification of the RFPM and pilot testing with 4 adolescents, we will test the reliability and validity of both the RFPM and food records when used by 60 adolescents (12 to 18 years of age). During one week, participants will use the RFPM and during another week they will use food records (the order will be balanced across participants). The accuracy of each method will be examined by comparing energy and nutrient intake (collectively referred to as food intake or FI) to three gold standards: 1) doubly labeled water or DLW (energy intake only, or EIDLW), 2) a laboratory-based test meal (FILaboratory), and 3) food intake during lunch in a school cafeteria (FISchool). User-satisfaction and participant burden will also be compared between methods, and a cost-effectiveness analysis will determine if and under what conditions one method is more cost-effective than the other.

ELIGIBILITY:
Inclusion Criteria:

* boy or girl of any race
* age 12 to 18 years, inclusive
* willing to use the RFPM for one week and pen-and-paper food records for one week
* willing to complete one laboratory-based food test during week 3
* willing to use the RFPM and food records during the laboratory-based test.

Exclusion Criteria:

-weight unstable (>1.1 pounds weight change in one week based on regressed daily body weights).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 50 adolescents will be recruited.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Doubly Labeled Water (DLW) | 2 weeks
  Doubly labeled water will be used to measure total daily energy expenditure (TEE) and Energy Intake.

SECONDARY OUTCOMES:
The Remote Food Photography Method (RFPM) | 7 days
  In brief, adolescents will be trained to use a Smartphone and the Food Image App to capture images of their food selection and plate waste and to send the data packets to Food Photo II via the wireless network.

OTHER OUTCOMES:
Pen-and-paper Food Records | 7 days
  Participants will be instructed how to keep a food record and estimate portion size during a session at the Center. Participants will also receive a packet containing the food protocol outline, food record form, guide to portion sizes, guidelines for description of foods, and tips for recording food intake. Participants will be instructed to record everything they eat or drink, recording the food item, portion size, time of consumption, and meal designation.

CONTACTS AND LOCATIONS:
Overall Officials: Corby K Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States